CLINICAL TRIAL: NCT01951274
Title: A Phase II Randomized, Double Blind, Parallel Group, Placebo-Controlled Dose Finding and Efficacy Study of VPD-737 in the Treatment of Subjects With Chronic Pruritus
Brief Title: VPD-737 for Treatment of Chronic Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCP 101
Record Dates: First submitted 2013-07-19; First posted 2013-09-26 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pruritus
MeSH Terms: interventions — serlopitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.25 mg VPD-737 (Experimental): 0.25 mg of VPD-737 daily by mouth for 42 days
  Interventions: Drug: VPD-737
- 1 mg VPD-737 (Experimental): 1 mg VPD-737 taken daily by mouth for 42 days
  Interventions: Drug: VPD-737
- 5 mg VPD-737 (Experimental): 5 mg tablets of VPD-737 to be taken daily by mouth for 42 days
  Interventions: Drug: VPD-737
- Placebo (Placebo Comparator): placebo tablets to be taken daily by mouth for 42 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VPD-737 — NK1 Receptor Antagonist
  Other Names: Serlopitant
  Arms: 0.25 mg VPD-737; 1 mg VPD-737; 5 mg VPD-737
Drug: Placebo
  Arms: Placebo

SUMMARY:
A study of a several doses of a novel treatment for chronic itch compared to placebo for patients whose condition has not responded to other treatments

DETAILED DESCRIPTION:
The sensation of itch is transmitted to the brain through the nervous system Several chemicals are involved in transmitting this signal This trial of VPD 737 is intended to treat this condition by blocking one of the chemicals involved in the transmission of the itch signal This is an oral drug administered once daily It has been used in other trials and has shown to be safe at the doses used in this trial The trial will involve once daily pills for 6 weeks. Subject will be asked to fill out questionnaires both electronically and on paper during the study period Patients will also be monitored for safety and will have blood taken for testing and several points during the trial Overall participation will last about 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic pruritus and unresponsive to current therapies

Exclusion Criteria:

* Have chronic liver or renal disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2014-12-02 (Actual); Study Completion 2014-12-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 6 weeks

SECONDARY OUTCOMES:
Verbal Response Scale | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Schnipper, MD, Study Director — Acting Chief Medical Officer, Tigercat Pharma, Inc.
Locations (25):
- United States (25):
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Stanford University, Medical Dermatology, Redwood City, California
  - UCSD Dermatology, San Diego, California
  - The Center for Clinical and Cosmetic Research, Aventura, Florida
  - Dermatology of Boca, Boca Raton, Florida
  - Skin Care Research, Boca Raton, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Advanced Medical Research, Inc., Atlanta, Georgia
  - Shideler Clinical Research Center, Carmel, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Grekin Skin Institue, Warren, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Quality Clinical Research Inc., Omaha, Nebraska
  - Comprehensive Clinical Research, Berlin, New Jersey
  - The Dermatology Group, P.C., Verona, New Jersey
  - Skin Search of Rochester, Inc., Rochester, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Baker Allergy, Asthma and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - Suzanne Bruce and Associates, P.A., Houston, Texas
  - Pfugerville Dermatology, Pflugerville, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - WestEnd Dermatology Associates, Richmond, Virginia
  - Marycliff Allergy Specialist, Spokane, Washington

REFERENCES:
- [Derived] Yosipovitch G, Stander S, Kerby MB, Larrick JW, Perlman AJ, Schnipper EF, Zhang X, Tang JY, Luger T, Steinhoff M. Serlopitant for the treatment of chronic pruritus: Results of a randomized, multicenter, placebo-controlled phase 2 clinical trial. J Am Acad Dermatol. 2018 May;78(5):882-891.e10. doi: 10.1016/j.jaad.2018.02.030. Epub 2018 Feb 17. PMID 29462657